CLINICAL TRIAL: NCT06563583
Title: Comparison of the Effectiveness of Self-Pressurizing Air-Q Intubating Laryngeal Airways Among Different Age Groups
Brief Title: Comparison of the Effectiveness of Air-Q SP Among Different Age Groups
Status: Completed | Type: Observational
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Zeynep Koc, principal investigator, Diskapi Yildirim Beyazit Education and Research Hospital
Other Study IDs: ZeynepKoc001
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Postoperative Complications; Sore-throat; Airway Complication of Anesthesia
Keywords: Air-Q SP İntubating Laryngeal Airway; oropharyngeal leak pressure; supraglottic airways
MeSH Terms: conditions — Postoperative Complications; Pharyngitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Group 1 will include patients aged 18-40 years.
  Interventions: Other: Group 1 will include patients aged 18-40 years
- Group 2: Group 2 will include patients aged 40-64 years.
  Interventions: Other: Group 2 will include patients aged 40-64 years
- Group 3: Group 3 will include patients aged 65-85 years.
  Interventions: Other: Group 3 will include patients aged 65-85 years

INTERVENTIONS:
Other: Group 1 will include patients aged 18-40 years — Group 1 will include patients aged 18-40 years.
  Groups: Group 1
Other: Group 2 will include patients aged 40-64 years — Group 2 will include patients aged 40-64 years, and finally.
  Groups: Group 2
Other: Group 3 will include patients aged 65-85 years — Group 3 will include patients aged 65-85 years.
  Groups: Group 3

SUMMARY:
Some previous studies have reported structural and physiological changes in the pharyngeal airway and UES with aging . It has been found that the shape and size of the pharyngeal airway in elderly individuals differ from those of young adults. This study aims to compare the effectiveness of the Air-Q laryngeal mask airway (LMA) across different age groups (young, middle-aged, and elderly patients) and to evaluate complications associated with supraglottic airways (SGA).

DETAILED DESCRIPTION:
"Supraglottic airway devices (SGA) used perioperatively are known to require lower anesthetic depth and result in fewer airway complications such as coughing and sore throat after awakening from anesthesia compared to endotracheal intubation. Due to these advantages, SGAs are particularly beneficial in elderly patients, as they experience a reduction in functional reserves, are more affected by cardiopulmonary diseases, and are more sensitive to anesthetic drugs

SGAs are inserted through the oral route, and the SGA cuff is placed between the base of the tongue, hypopharynx, and upper esophageal sphincter (UES) to provide proper ventilation. Some previous studies have reported structural and physiological changes in the pharyngeal airway and UES with aging . It has been found that the shape and size of the pharyngeal airway in elderly individuals differ from those of young adults. Additionally, there are changes in the function and structure of the UES with age. These age-related changes may affect the performance of SGAs in the elderly population.

Recently, SGAs that do not require manual cuff inflation have been used more frequently in various clinical settings due to the advantages of eliminating the need for manual cuff inflation and cuff pressure monitoring. The Air-Q is connected to an airway tube through a communication port that allows for self-regulation of cuff pressure in response to airway pressure."

ELIGIBILITY:
Inclusion Criteria:

* 18-85 year-old patients
* American Society of Anesthesiologist Physical Status classification I-III,
* Undergoing an elective operation under general anesthesia in our hospital

Exclusion Criteria:

* Predicted difficult airway (Mallampati class 4, mouth opening < 3 cm, or thyromental distance < 6 cm)
* body mass index (BMI) > 40 kg/m2
* Patients with a high risk of aspiration (e.g., history of gastrectomy, gastroesophageal reflux disease, or hiatal hernia),
* Unstable vital signs,
* Cervical spine problems, Respiratory complications (e.g. recent pneumonia).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective surgery under general anesthesia with the use of an SP Air-Q.
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2024-09-02 (Actual); Primary Completion 2024-11-07 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Measurement of oropharyngeal leak pressure (OLP) | One minute after successful LMA placement
  One minute after successful LMA placement and fixation, oropharyngeal leak pressure (OLP) will be measured by setting the adjustable pressure limiting valve (APL) to 40 mmHg and maintaining a fresh gas flow of 3 L/min. The OLP will be recorded as the pressure at which an audible leak sound is heard from the mouth.

SECONDARY OUTCOMES:
SP Air-Q insertion time | 3 minutes after induction of anesthesia
  Successful LMA placement will be confirmed by visualizing a square waveform on the ventilator and observing chest wall movement.
ease of LMA placement | 3 minutes after induction of anesthesia
  The ease of LMA placement will be scored by the anesthesiologist on a scale from 1 to 4 (1: Successful on the first attempt with no resistance from the tissues; 2: Successful on the first attempt but with some tissue resistance during placement; 3: Moderate tissue resistance; 4: Failure to place the LMA).
maneuvers required for successful ventilation | 3 minutes after induction of anesthesia
  It will be recorded whether any further maneuvers are required: Gentle pushing or pulling of the LMA to adjust its depth, jaw-thrust maneuver, and flexion or extension of the head.
fiberoptic view grading | 3 minutes after induction of anesthesia
  The Brimacombe score will be used to evaluate the view obtained with fiberoptic bronchoscopy. 1: Vocal cords are not visible; 2: Vocal cords and anterior epiglottis are visible; 3: Vocal cords and posterior epiglottis are visible; 4: Vocal cords are visible.
Complications during SP_Air-Q removal (emerge) | One minute after SP Air-Q removal
  such as breath-holding during emergence, airway obstruction, coughing, hypoxia (SpO2 < 90%), vomiting, lip-tongue-teeth trauma, and bleeding, will be recorded
sore throat | 1-24 hours postoperatively
  Postoperative complication
dysphonia | 1-24 hours postpoeratively
  Postoperative complication

CONTACTS AND LOCATIONS:
Locations (1):
- Zeynep Koç, Yenimahalle, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lee JS, Kim DH, Choi SH, Ha SH, Kim S, Kim MS. Prospective, Randomized Comparison of the i-gel and the Self-Pressurized air-Q Intubating Laryngeal Airway in Elderly Anesthetized Patients. Anesth Analg. 2020 Feb;130(2):480-487. doi: 10.1213/ANE.0000000000003849. PMID 30320644
- [Result] Kim EM, Kim MS, Koo BN, Lee JR, Lee YS, Lee JH. Clinical efficacy of the classic laryngeal mask airway in elderly patients: a comparison with young adult patients. Korean J Anesthesiol. 2015 Dec;68(6):568-74. doi: 10.4097/kjae.2015.68.6.568. Epub 2015 Nov 25. PMID 26634080
- [Result] Kim MH, Lee JH, Choi YS, Park S, Shin S. Comparison of the laryngeal mask airway supreme and the i-gel in paralysed elderly patients: A randomised controlled trial. Eur J Anaesthesiol. 2018 Aug;35(8):598-604. doi: 10.1097/EJA.0000000000000700. PMID 28857785